CLINICAL TRIAL: NCT04981444
Title: Optimization of an Automated Ultrasound Cardiac Guidance Tool
Status: Completed | Type: Observational
Sponsor: UltraSight (Industry)
Responsible Party: Sponsor
Other Study IDs: 002-20
Record Dates: First submitted 2021-07-04; First posted 2021-07-29 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-07

CONDITIONS: Ultrasound Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Open-label, single-arm, prospective study. Subjects will undergo one session of 2D Transthoracic Echocardiogram (2D-TTE) ultrasound. The ultrasound will be performed by a trained sonographer.

DETAILED DESCRIPTION:
The study will use a commercially available handheld imaging device (Philips Lumify transducer).

Primary Objective:

To acquire images of multiple transducer position, trajectories, and views, at different acoustic windows for capturing images and location relative to body and probe positions.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and above.
2. Patients able to understand, read and sign the informed consent
3. Patient willing to answer a short questionnaire

Exclusion Criteria:

1. Pregnancy(females of childbearing potential will be tested with a urine pregnancy test prior to their inclusion in the study)
2. Not willing or not able to sign an inform consent
3. Physical limitation to maneuvering the probe on the body
4. Unable to lie flat for study
5. Patients experiencing a known or suspected acute cardiac event
6. Patients with severe chest wall abnormalities
7. Patients who have undergone pneumonectomy
8. Patients whose anatomy does not lend itself to echocardiography

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Up to 75 cardiac patients will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2021-07-22 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2022-09-23 (Actual)

PRIMARY OUTCOMES:
ACCURACY- Optimization of an automated ultrasound cardiac guidance tool. | 1 year
  To acquire images from different transducer positions, trajectories, and views, at different acoustic windows for capturing images and location relative to body and probe.
  This study is designed to capture data for the training of the UltraSight Guidance software AI models. The obtained data will not be anlyzed for statistical purposes but will only be used for the algorithm development based on the technician movements recording, with no reference to images quality or medical utilization.

CONTACTS AND LOCATIONS:
Overall Officials: Praveen Mehrotra, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No